CLINICAL TRIAL: NCT02358980
Title: KIDNEY THERAPY FOR FREE LIGHT CHAIN REMOVAL IN PATIENTS WITH MULTIPLE MYELOMA & CAST NEPHROPATHY
Acronym: KEEPER
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 73/2014
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma; Cast Nephropathy; Acute Kidney Injury
Keywords: Multiple Myeloma; Cast Nephropathy; Acute kidney injury; KIDNEY THERAPY; HFR
MeSH Terms: conditions — Multiple Myeloma; Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study group: Participants will receive FLC removal HD undertaken using an extended dialysis schedule on KIDNEY therapy system. Treatments (4 hours each) were carried out for 8 consecutive days and then every other day.
  Interventions: Device: KIDNEY therapy

INTERVENTIONS:
Device: KIDNEY therapy

SUMMARY:
Hypothesis: Free light chain (FLC) removal haemodialysis will increase the rate of renal recovery in patients with cast nephropathy, severe renal failure and de novo multiple myeloma.

This study will evaluate patients with multiple myeloma and severe renal failure treated with KIDNEY Therapy (previously called SUPRA HFR) to remove free light chains.

DETAILED DESCRIPTION:
This is an observational study performed to investigate the clinical benefit of FLC removal by KIDNEY therapy system in patients with cast nephropathy, dialysis dependent renal failure and de novo multiple myeloma. Recruitment commenced in July 2014, in total 20 patients will be recruited. Participants will be treated with, KIDNEY therapy system (Bellco Mirandola, Modena, Italy) . The KIDNEY system is a kind of haemodiafiltration that utilizes separated convection, diffusion and adsorption. The sorbent cartridge has a high affinity for FLC (both κ and λ) but is able to re-infuse albumin, avoiding the need for albumin perfusions. The KIDNEY therapy will be undertaken over an intensive treatment schedule. The primary outcome for the study is independence of dialysis in 3 month. Secondary outcomes are: duration dialysis, reduction of serum FLC levels, myeloma response and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Dialysis dependent acute renal failure
* Fulfils diagnostic criteria for the diagnosis of symptomatic de novo multiple myeloma
* Abnormal serum FLC ratio and a sFLC concentration > 500 mg/L
* Myeloma kidney demonstrated on a renal biopsy (cast nephropathy)
* Ability to give informed consent to partake in study
* Commencement of study within 10 days of presenting to enrolling unit

Exclusion Criteria:

* Known advanced chronic renal failure (CKD stage IV 4-5; eGFR <30mls/min/1.73m2) or evidence of significant chronic damage on renal biopsy
* Amyloidosis or light chain deposition disease on renal biopsy
* Previous treatment of multiple myeloma with chemotherapy
* Haemodynamic instability that precludes unsupported dialysis renal replacement therapy
* Significant cardiac disease
* Active uncontrolled infection
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cast nephropathy, dialysis dependent renal failure and de novo multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Independence of haemodialysis at 3 months from enrollment | 3 months from enrollment

SECONDARY OUTCOMES:
Efficency of KIDNEY therapy system with respect to reduced sFLC levels | 21 days from enrollment
Duration of HD from renal recover | 3 months from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology and Dialysis Unit ASMN IRCCS, Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Background] Winearls CG. Acute myeloma kidney. Kidney Int. 1995 Oct;48(4):1347-61. doi: 10.1038/ki.1995.421. No abstract available. PMID 8569099
- [Background] Haubitz M, Peest D. Myeloma--new approaches to combined nephrological-haematological management. Nephrol Dial Transplant. 2006 Mar;21(3):582-90. doi: 10.1093/ndt/gfi318. Epub 2006 Jan 5. No abstract available. PMID 16396976
- [Background] Hutchison CA, Cockwell P, Reid S, Chandler K, Mead GP, Harrison J, Hattersley J, Evans ND, Chappell MJ, Cook M, Goehl H, Storr M, Bradwell AR. Efficient removal of immunoglobulin free light chains by hemodialysis for multiple myeloma: in vitro and in vivo studies. J Am Soc Nephrol. 2007 Mar;18(3):886-95. doi: 10.1681/ASN.2006080821. Epub 2007 Jan 17. PMID 17229909
- [Background] Hutchison CA, Blade J, Cockwell P, Cook M, Drayson M, Fermand JP, Kastritis E, Kyle R, Leung N, Pasquali S, Winearls C; International Kidney and Monoclonal Gammopathy Research Group. Novel approaches for reducing free light chains in patients with myeloma kidney. Nat Rev Nephrol. 2012 Feb 21;8(4):234-43. doi: 10.1038/nrneph.2012.14. PMID 22349488
- [Background] Testa A, Dejoie T, Lecarrer D, Wratten M, Sereni L, Renaux JL. Reduction of free immunoglobulin light chains using adsorption properties of hemodiafiltration with endogenous reinfusion. Blood Purif. 2010;30(1):34-6. doi: 10.1159/000316684. Epub 2010 Jun 24. PMID 20588010
- [Background] Pasquali S, Iannuzzella F, Corradini M, Mattei S, Bovino A, Stefani A, Palladino G, Caiazzo M. A novel option for reducing free light chains in myeloma kidney: supra-hemodiafiltration with endogenous reinfusion (HFR). J Nephrol. 2015 Apr;28(2):251-4. doi: 10.1007/s40620-014-0130-8. Epub 2014 Aug 23. PMID 25149172